CLINICAL TRIAL: NCT05233618
Title: Phase I Study of Tagraxofusp for Post-Transplant Maintenance for Patients With CD 123+ Acute Myeloid Leukemia, Myelodysplastic Syndrome, Myelofibrosis and Chronic Myelomonocytic Leukemia
Brief Title: Study of Tagraxofusp for Post-Transplant Maintenance for Patients With CD 123+ AML, MDS, MF and CMML (HSCT 002)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Karen Ballen, MD (Other)
Responsible Party: Sponsor-Investigator, Karen Ballen, MD, Chief of the Hematology/Oncology Division and the Medical Director of the Stem Cell Transplant Program, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR210434
Record Dates: First submitted 2022-01-19; First posted 2022-02-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Myelofibrosis; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia
Keywords: Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — tagraxofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tagraxofusp (escalating doses) (Experimental): IV tagraxofusp on days 1-3 of cycles 1-4 and days 1-2 of additional cycles for up to 9 cycles (some participants could receive more if considered in their best interest)
  Interventions: Drug: Tagraxofusp

INTERVENTIONS:
Drug: Tagraxofusp — inpatient on days 1-3 of cycles 1-4 and days 1-2 of additional cycles
  Other Names: SL-701, Elzonris

SUMMARY:
In this study, tagraxofusp (Tag) is given to patients with CD 123+ myelofibrosis (MF), chronic myelomonocytic leukemia (CMML), and acute myeloid leukemia (AML) after allogeneic stem cell transplant (HCT) to help prevent relapse. Patients will receive up to about 9 cycles of treatment with Tag and have a bone marrow biopsy after cycle 4 and about 1 year after HCT.

DETAILED DESCRIPTION:
Relapsed disease is the primary cause of treatment failure after hematopoietic cell transplant (HCT). In this study, patients are given increasing levels of tagraxofusp (Tag) to evaluate the safety of each dose. Participants will start treatment with Tag starting between 60 and 120 days following HCT. Tag will be given by IV over about 15 minutes on days 1 through 3 of cycles 1-4 of treatment (28 day cycles) and then on days 1 and 2 of subsequent cycles, for up to 9 cycles or until disease progression or if you have a bad side effect. In the first cycle, Tag will be given while participants are inpatient. In all other cycles, Tag will be given outpatient and participants will be observed for 4 hours following each infusion. After about 4 cycles of treatment and again about 1 year after HCT, participants will have a bone marrow biopsy and also take a questionnaire about their quality of life. During the study, participants will have their blood checked regularly to monitor for side effects.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is ≥18 years old and ≤ 75 years old.
2. The patient has a life expectancy of >6 months.
3. The patient has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2.
4. The patient has adequate baseline organ function, including cardiac, renal, and hepatic function within 28 days of start of therapy:

   * Left ventricular ejection fraction (LVEF) ≥ 50% as measured by multigated acquisition scan (MUGA) or 2-dimensional (2-D) echocardiogram (ECHO) and no clinically significant abnormalities on a 12-lead electrocardiogram (ECG)
   * Serum Creatinine ≤ 1.5 mg/dL
   * Bilirubin ≤1.5 mg/dL
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 times the upper limit of normal (ULN)
   * Absolute neutrophil count (ANC) ≥0.5 × 10⁹/L
   * Platelets ≥ 80,000/mm^3
   * Serum albumin ≥3.2 (note that albumin infusions are not permitted in order to enable eligibility)
5. Patient meets the 2016 WHO diagnostic criteria for MF, is CD 123+, and has an IPSS/DIPSS/DIPSS-plus intermediate-1 with anemia (Hb < 10g/dl), splenomegaly (> 12 cm), leukocytosis (WBC > 25K) intermediate-2 or high-risk disease pre transplant.

   Or

   Patient has a 2016 WHO-defined diagnosis of CMML (persistent monocytosis ≥1 × 10⁹/L for at least 3 months, with other causes excluded, and monocytes ≥10% of WBC in peripheral blood, no criteria and no previous history of CML, ET, PV, and acute promyelocytic leukemia) pre transplant and is CD123+

   Or

   Patient has 2016 WHO-defined CMML-1 (2-4% blasts in peripheral blood and/or 5-9% blasts in bone marrow) and CMML-2 (5-19% blasts in peripheral blood and/or 10-19% blasts in bone marrow, and/or presence of Auer rods) pre transplant and is CD 123+

   Or

   Patient has CD 123+ AML in morphologic remission pre transplant

   Or

   Patient has Intermediate or high risk MDS by IPSS-R or moderate or high risk by IPSS-M pre transplant and has had no morphologic progression of disease post-transplant.

   Receipt of first allogeneic stem cell transplant (related, unrelated, haploidentical or cord blood) 60-120 days prior to study registration
6. Patient is in morphologic remission according to bone marrow biopsy completed within 30 days prior to planned start of study treatment
7. Provision of signed and dated informed consent form
8. Stated willingness to comply with all study procedures and availability for the duration of the study
9. For females and males of reproductive potential: agreement to use adequate contraception for at least one month prior to screening, during study participation and for an additional one week after the end of study drug administration. Other (non-study) medications may require participants to use adequate contraception for longer.
10. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner. Other (non-study) medications may require participants to use adequate contraception for longer.
11. Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

1. Treatment with any disease-related therapy, including radiation therapy or investigational agent, within 14 days of study entry
2. Previous treatment with tagraxofusp or known hypersensitivity to any components of the drug product
3. Active malignancy and/or cancer history (excluding myeloproliferative disorders and concomitant myeloid malignancies as specified in the inclusion criteria) that can confound the assessment of the study endpoints. Patients with a past cancer history (within 2 years of entry) and/or ongoing active malignancy or substantial potential for recurrence must be discussed with the Sponsor before study entry. Patients with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including superficial bladder cancer), cervical intraepithelial neoplasia, or organ-confined prostate cancer with no evidence of progressive disease.
4. Known active or suspected disease involvement of the central nervous system (CNS)
5. Receiving > 10 mg prednisone daily for GVHD
6. Overall Grade 2 or greater acute GVHD (per Magic criteria) at time of registration
7. Pregnant or breast feeding
8. Requirement of supplemental oxygen
9. Clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction or stroke within 6 months of study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication)
10. Uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study
11. Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements
12. Known positive status for human immunodeficiency virus or active or chronic Hepatitis B or Hepatitis C
13. Receiving treatment for known or suspected fungal infection (prophylaxis is acceptable)
14. Known positive SARS-COV-2 test within 3 weeks of study entry. Exception: Tests that reflect past, resolved infection where the patient is determined to NOT be infectious, according to an infectious disease specialist, do not exclude the patient from participation.
15. Pedal edema ≥ grade 2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of grade ≥ 3 adverse events | Through about 30 days following last infusion of tagraxofusp
  Severity is based upon CTCAE v5 criteria.
Dose limiting toxicities | During cycles 1 and 2 (each cycle is 28 days) of study treatment for each participant
  Frequencies of certain, more severe, types of side effects from the study drug
Percent of planned tagraxofusp dose received | Through cycle 4 (each cycle is 28 days) of study treatment for each participant
  During cycles 1-4 only

SECONDARY OUTCOMES:
Time from HCT to relapse and death or last contact. | Participants will be followed through 2 years after date of HCT
  Duration
Frequency and severity of acute GVHD grades II-IV and chronic GVHD | Participants will be followed through 2 years after date of HCT
  Mild, moderate or severe per Magic criteria

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ballen, Principal Investigator — UVA
Locations (2):
- United States (2):
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No